CLINICAL TRIAL: NCT00981604
Title: Single Incision Versus Laparoscopic Cholecystectomy
Brief Title: Single Incision Laparoscopic Surgery (SILS) Versus Laparoscopic Cholecystectomy
Acronym: SILS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Shawn St. Peter, MD, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09 07 132
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Cholelithiasis; Biliary Dyskinesia
Keywords: SILS; Laparoscopic Cholecystectomy; Children
MeSH Terms: conditions — Cholelithiasis; Biliary Dyskinesia | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SILS Cholecystectomy (Active Comparator): Single Incision Laparoscopic Cholecystectomy
  Interventions: Procedure: SILS
- Standard Laparoscopic Cholecystectomy (Active Comparator): 4 port laparoscopic cholecystectomy
  Interventions: Procedure: Standard Laparoscopic Cholecystectomy

INTERVENTIONS:
Procedure: SILS — Single Incision Laparoscopic Cholecystectomy
  Arms: SILS Cholecystectomy
Procedure: Standard Laparoscopic Cholecystectomy — 4 port technique
  Other Names: Laparoscopic Cholecystectomy
  Arms: Standard Laparoscopic Cholecystectomy

SUMMARY:
Prospective randomized trial of single incision versus standard 4 port laparoscopic cholecystectomy. Hypothesis is that the operative time will be longer with single incision.

DETAILED DESCRIPTION:
This will be a prospective, randomized clinical trial involving patients who present to the hospital with an indication for cholecystectomy. We will offer enrollment to several institutions provided they receive institutional approval.

This will be a definitive trial design. Based on our operative times with SILS compared with our recent experience in standard laparoscopy, a sample size of 60 patients will give us a power of 0.8 with an α of 0.05.

After the procedure, both groups will be managed in the same manner per routine care. They will be discharged when tolerating a regular diet and their pain is well-controlled on oral pain medication.

ELIGIBILITY:
Inclusion Criteria:

* Need for cholecystectomy

Exclusion Criteria:

* Need for cholangiogram

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Operative Time | 1 day

SECONDARY OUTCOMES:
Operative complications | 2 weeks
length of hospitalization | 1 week
doses of analgesics | 1 week
hospital/operation charges | 1 week
surgeon perception of difficulty | 1 day
cosmetic scores | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Ostlie, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

REFERENCES:
- [Derived] Ostlie DJ, Juang OO, Iqbal CW, Sharp SW, Snyder CL, Andrews WS, Sharp RJ, Holcomb GW 3rd, St Peter SD. Single incision versus standard 4-port laparoscopic cholecystectomy: a prospective randomized trial. J Pediatr Surg. 2013 Jan;48(1):209-14. doi: 10.1016/j.jpedsurg.2012.10.039. PMID 23331817